CLINICAL TRIAL: NCT07340411
Title: Effect of Chinese Herbal Medicine Nasal Irrigation on the Postoperative Care of Chronic Rhinosinusitis
Acronym: Breeze Clear
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Rong-San Jiang, visiting doctor, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CF23171A; TCVGH-1137302C (Other Grant/Funding Number: Taichung Veterans General Hospital)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Chronic Rhinosinusitis; Postoperative Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese herbal medicine (Experimental): In the Chinese herbal medicine group, Chinese herbal medicine nasal irrigant was first prepared by mixing a pack of 2 gram of SHIN YI CHING FEY TANG, 0.5 gram of chrysanthemum, and 0.125 gram of Borneo camphor powder with 240mL of sterile water in the container of the irrigator. Nasal irrigation was performed by using a NeilMed® SINUS RINSE™ Squeeze Bottle (NeilMed Pharmaceuticals, Inc., Santa Rosa, CA ). When irrigating the nose, patients irrigated both of their nasal cavities each with 120 mL of solutions twice a day. Patients performed nasal irrigations for 2 months.
  Interventions: Drug: Chinese herbal medicine Powder
- Saline (Placebo Comparator): In the saline group, the normal saline solution was prepared by mixing 1 pack of 2.16 gram salt powder with 240mL of sterile water in the container of the irrigator. Nasal irrigation was performed by using a NeilMed® SINUS RINSE™ Squeeze Bottle (NeilMed Pharmaceuticals, Inc., Santa Rosa, CA ). When irrigating the nose, patients irrigated both of their nasal cavities each with 120 mL of solutions twice a day. Patients performed nasal irrigations for 2 months.
  Interventions: Drug: Salt Powder

INTERVENTIONS:
Drug: Chinese herbal medicine Powder — The bilateral nasal cavity was irrigated by using a NeilMed® SINUS RINSE™ Squeeze Bottle containing 240ml of Chinese herbal medicine solution twice a day for 2 months.
  Other Names: 2 gram of SHIN YI CHING FEY TANG, 0.5 gram of chrysanthemum, and 0.125 gram of Borneo camphor
  Arms: Chinese herbal medicine
Drug: Salt Powder — The bilateral nasal cavity was irrigated by using a NeilMed® SINUS RINSE™ Squeeze Bottle containing 240ml of of normal saline twice a day for 2 months.
  Arms: Saline

SUMMARY:
Investigators tried to evaluate the efficacy and safety of Chinese herbal medicine nasal irrigation as an adjuvant therapy after FESS.

DETAILED DESCRIPTION:
In this study, patients with chronic rhinosinusitis who received FESS were recruited and randomly assigned to 2 groups at one month post-surgery. Patients in the xylitol group received 240ml of Chinese herbal medicine nasal irrigation daily for 2 months, and those in the normal saline (NS) group received 240ml of NS nasal irrigation daily for 2 months. Before FESS as well as before and after nasal irrigation, sino-nasal symptoms were assessed by a 22-item Sino-Nasal Outcome Test questionnaire and patients received endoscopic examination, nasal function tests, cytokine measurement of nasal irrigant, and bacterial culture from the middle meatus. The safety of nasal irrigation was assessed by self-reported adverse events, and blood test. This study tried to evaluate the efficacy and safety of Chinese herbal medicine nasal irrigation as an adjuvant therapy after FESS.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with chronic rhinosinusitis who failed medical treatment 2.Patients underwent bilateral primary functional endoscopic sinus surgery.

Exclusion Criteria:

* 1. Patients with a history of immunodeficiency 2.Patients with a history of sinus surgery 3.Patients who receiving antibiotic treatment within a week before functional endoscopic sinus surgery 4.Patients with a pathological diagnosis of fungal sinusitis 5.Patients with a pathological diagnosis of sinonasal tumor

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Taiwanese version of the 22-item Sino-Nasal Outcome Test | From before operation to 3 months after surgery
  The Taiwanese version of the 22-item Sino-Nasal Outcome Test contains 22 items of symptoms and social/emotional consequences from nasal disorder. Patients are asked to rate their problems based on how they have been over the past two weeks. Each item is graded from 0 (no problem) to 5 (as bad as it can be) according to its severity and frequency.
Self-reported adverse events | From before nasal irrigation to after 2-month nasal irrigation
  Any adverse events occurring during the 2 months period of nasal irrigation

SECONDARY OUTCOMES:
Change of the second minimal cross-sectional area of the nasal cavity | From before operation to 3 months after surgery
  The second minimal cross-sectional area of the nasal cavity was measured by acoustic rhinometry.
Change of endoscopic score | From before operation to 3 months after surgery
  The endoscopic appearances were categorized into polyps (0: no polyps; 1: polyps present within the middle meatus; 2: polyps beyond the middle meatus); nasal secretion (0: no secretion; 1: clear, thin secretion; 2: thick, purulent secretion); mucosal edema; scarring; crusting; (0: absent; 1: mild; 2: severe). The score ranged from 0 to 20 for both nostrils together.
Change of saccharine transit time | From before operation to 3 months after surgery
  The saccharine transit test involved placing saccharine granules under the head of the inferior turbinate in the more severely affected nostril. The time interval (minute) between placement of saccharine granules and sensation of sweetness in the throat was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Rong-San Jiang, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Outcome measures
Supporting Information: Study Protocol
Time Frame: 2 years after the end of the study
Access Criteria: Study Data/Document can be requested from the PI.
URL: https://www.vghtc.gov.tw/